CLINICAL TRIAL: NCT04894110
Title: A Phase 1, Prospective, Multi-Center, Open-Label, Dose-Escalation Study to Assess the Safety, and Tolerability of EO2002 with and Without Endothelial Brushing or Descemet Stripping in the Treatment of Corneal Edema (EMME-001)
Brief Title: Study of Safety and Tolerability of EO2002 in the Treatment of Corneal Edema
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emmecell (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EMME-001
Record Dates: First submitted 2021-05-11; First posted 2021-05-20 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Corneal Edema; Corneal Endothelial Dysfunction; Corneal Endothelial Dystrophy; Fuchs Dystrophy; Fuchs Endothelial Corneal Dystrophy; Pseudophakic Bullous Keratopathy; Bullous Keratopathy; Endothelial Dysfunction; Moderate Corneal Endothelial Decompensation
MeSH Terms: conditions — Corneal Edema; Corneal Dystrophy, Posterior Polymorphous, 1; Fuchs' Endothelial Dystrophy

STUDY DESIGN:
Intervention Model Description: Group 1: Open-Label, Dose-Escalation Study Group 2: Randomized, double masked
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- EO2002 treatment - Group 1 (Experimental)
  Interventions: Biological: EO2002
- EO2002 treatment - Group 2 - low dose (Active Comparator)
  Interventions: Biological: EO2002 low dose
- EO2002 treatment - Group 2 - mid dose (Active Comparator)
  Interventions: Biological: EO2002 mid dose
- EO2002 treatment - Group 2 - high dose (Active Comparator)
  Interventions: Biological: EO2002 high dose

INTERVENTIONS:
Biological: EO2002 — EO2002 (magnetic human corneal endothelial cells [HCECs]) with and without endothelial brushing (EB) or Descemet Stripping (DS)
  Arms: EO2002 treatment - Group 1
Biological: EO2002 low dose — Low dose of EO2002 (magnetic human corneal endothelial cells)
  Arms: EO2002 treatment - Group 2 - low dose
Biological: EO2002 mid dose — Mid dose of EO2002 (magnetic human corneal endothelial cells)
  Arms: EO2002 treatment - Group 2 - mid dose
Biological: EO2002 high dose — High dose of EO2002 (magnetic human corneal endothelial cells)
  Arms: EO2002 treatment - Group 2 - high dose

SUMMARY:
Corneal edema is the most common indication for corneal transplantation, accounting for approximately 70% of penetrating keratoplasty (PK), and 100% of endothelial keratoplasty (EK) procedures annually. There is currently no disease-modifying treatment for corneal edema. Topical treatments like hypertonic saline are not effective on a long-term basis. For those with advanced disease, where edema and vision loss are not controlled by topical treatment, the only option is a corneal transplant. A potential approach to avoidance of the risks of corneal transplantation is to inject cultured human corneal endothelial cells (HCECs) into the anterior chamber of the eye. This approach may avoid surgery by re-populating the inner most aspect of the cornea with functioning endothelial cells. Emmecell has developed a treatment based on technology integrating biocompatible magnetic nanoparticles with cultured HCECs to treat corneal edema in a minimally invasive way. The primary objective of this phase 1, prospective, multi-center, open-label, dose-escalation study is to evaluate the safety and tolerability of 3 doses of EO2002 with and without endothelial brushing (EB) or Descemet Stripping (DS) in eyes with corneal edema secondary to corneal endothelial dysfunction that qualify for surgery involving full-thickness corneal transplantation or EK.

DETAILED DESCRIPTION:
The study is designed to occur in 2 groups. The objective with the first group is to preliminarily evaluate the safety of 4 escalating doses. The purpose of the second group is to gather additional safety information on the 3 highest doses when administered according to a randomized schedule and evaluated by masked observers.

Group 1: Phase 1 prospective, multi-center, open-label, dose-escalation study designed to evaluate the safety and tolerability of EO2002 with and without endothelial brushing (EB) or Descemet Stripping (DS) in eyes with corneal edema secondary to corneal endothelial dysfunction that qualify for surgery involving full-thickness corneal transplantation or EK. Four doses will be studied in approximately 21 study participants that meet the inclusion/exclusion criteria. Safety and tolerability will be the primary focus for 26 weeks following treatment with EO2002.

Group 2: The three highest doses will be administered to up to 21 subjects in a randomized, double-masked design.

ELIGIBILITY:
Inclusion Criteria:

All ocular criteria apply to study eye unless otherwise noted.

1. Age ≥ 21 years.
2. Phakic or Pseudophakic with a posterior chamber intraocular lens
3. Symptomatic corneal edema associated with endothelial dysfunction which may be secondary to Fuchs corneal dystrophy or pseudophakic bullous keratopathy.

Exclusion Criteria:

All ocular criteria apply to study eye unless otherwise noted.

1. Other corneal disease
2. Anterior chamber intraocular lens, Sutured or scleral-fixated intraocular lens.
3. Macular disease that in the investigator and/or sponsor's opinion would limit the ability of the subject to demonstrate improvement in BCVA.
4. History of refractive surgery.
5. Descemet membrane detachment.
6. History of uveitis or other ocular inflammatory disease.
7. History of incisional glaucoma surgery (e.g.,trabeculectomy, glaucoma drainage implant).
8. Intraocular pressure >21 or <7 mm Hg
9. Prior incisional eye surgery within 3 months prior to study treatment or penetrating or endothelial keratoplasty.
10. History of ocular neoplasm.
11. ETDRS BCVA in the fellow eye is worse than 35 letters (Snellen equivalent of 20/200).
12. Female who is pregnant, nursing, or planning to become pregnant, or who is of childbearing potential and not using a reliable means of contraception during the study.
13. Subject is currently participating in or has participated within the last 3 months in any other clinical trial of an investigational drug by ocular or systemic administration.
14. Any concomitant medical or psychological condition that could interfere with study participation or is otherwise not suitable for entry into the study in the opinion of the investigator.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-06-22 (Actual); Primary Completion 2024-10-03 (Actual); Study Completion 2024-10-03 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability of EO2002] | 26 Weeks
  Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability of EO2002 (+/- EB or Descemet Stripping)] in subjects with corneal edema at week 26.

SECONDARY OUTCOMES:
Effect of EO2002 (+/-EB or DS) on corneal thickness | 26 Weeks
  Evaluate the effect of a single injection of EO2002 (+/-EB or DS) on corneal thickness as determined by pachymetry
Effect of EO2002 (+/-EB or DS) on best corrected visual acuity (BCVA). | 26 Weeks
  Evaluate the effect of a single injection of EO2002 (+/-EB or DS) on best corrected visual acuity (BCVA) as determined by ETDRS letter score.

CONTACTS AND LOCATIONS:
Overall Officials: Noelia Kunzevitzky, Study Director — Emmecell
Locations (8):
- United States (8):
  - Los Angeles Location, Greater Los Angeles, California
  - San Diego Location, San Diego, California
  - Miami Location, Miami, Florida
  - Palm Beach Gardens Location, Palm Beach Gardens, Florida
  - Atlanta Location, Atlanta, Georgia
  - Des Moines Location, Des Moines, Iowa
  - Kansas City Location, Overland Park, Kansas
  - Grand Rapids Location, Grand Rapids, Michigan

IPD SHARING:
Plan to Share IPD: No